CLINICAL TRIAL: NCT03865342
Title: Prevention of Diabetes Using Mobile-enabled, Virtual Delivery of the National Diabetes Prevention (DPP) Program: a Randomized Trial
Brief Title: Prevention of Diabetes Using Mobile-enabled, Virtual Delivery of the National Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Collaborators: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 695755-6
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: PreDiabetes
Keywords: mHealth; Diabetes Prevention Program; weight loss; body weight; behavioral interventions
MeSH Terms: conditions — Prediabetic State; Weight Loss; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noom Coach DPP (Experimental): Individuals will receive special instructions on how to use the app and will self-monitor their weight, exercise and receive daily DPP core content through the app over 16 weeks plus guidance from a coach, and will thereafter receive post-core DPP content up to 52 weeks.
  Interventions: Behavioral: Noom Coach DPP
- Usual Care (No Intervention): The control group will be a "usual care" condition in which participants are free to seek any assistance for their medical care during the study period plus a paper version of the DPP curriculum.

INTERVENTIONS:
Behavioral: Noom Coach DPP — Subjects receiving the smartphone app will receive the DPP core curriculum for 16 weeks and then the post-core curriculum for 36 weeks through the app. The Noom mobile app allows secure patient monitoring through a participant dashboard that the coach can use to increase patient adherence and motivation to achieve DPP goals. The participant can log their food intake, weight, steps, exercise, in addition to participating in the DPP group interaction through the application.
  Arms: Noom Coach DPP

SUMMARY:
This study will test the weight loss efficacy of a mobile diabetes prevention program intervention. Half of the sample of prediabetic adults will receive the virtual DPP and half will receive usual medical care.

DETAILED DESCRIPTION:
There were 84.1 million people with pre-diabetes, 30.3 million people with diagnosed and 7.2 million with undiagnosed diabetes in the United States in 2015, and nearly 2 million are diagnosed with it every year. By 2050, the CDC estimates that 1 in every 3 people globally will have diabetes, a leading cause of death and disability.

The primary goal of this study is to evaluate the efficacy of the Noom Coach Diabetes Prevention Program mobile platform versus usual medical care. The best intervention to date for prediabetes is the Centers for Disease Control and Prevention's Diabetes Prevention Program, yet there is limited research investigating a mobile-based delivery of the DPP. Pre-diabetes is often discovered during routine medical visitation/annual screening (usual care), but face-to-face time with clinicians is often limited. Exploring novel ways, such as mHealth interventions to empower patients to pursue lifestyle change and prevent or delay diabetes onset is critical to addressing the growing diabetes epidemic.

ELIGIBILITY:
Inclusion criteria:

* English-speaking
* 18 years of age and older
* Referral from the patient's physician
* Hemoglobin A1C: 5.7 - 6.4 within the 3 months prior to enrollment
* Own a smartphone (Apple or Android)

Exclusion criteria:

* Recent weight loss (by patient report, >5 lbs in the 6 months preceding enrollment visit)
* previous diagnosis of type 1 or type 2 diabetes
* serious or persistent mental illnesses
* more than 72 hours of hospitalization in the last 30 days
* Enrollment in a structured weight-loss program currently or within the 1 month preceding study enrollment
* Pregnant
* Currently nursing
* Have given birth within the past 3 months
* Has been discouraged by a physician to enroll in a DPP program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline, 6, and 12 months
  Body weight recorded during follow-up appointments at the medical clinic.

SECONDARY OUTCOMES:
Change in hemoglobin A1c | Baseline, 6, and 12 months
  Hemoglobin A1c measured during follow-up appointments at the medical clinic.

OTHER OUTCOMES:
Change in work productivity | Baseline, 6, and 12 months
  Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI)
  1. Are you currently employed (working for pay)?
  2. During the past seven days, how many hours did you miss from work because of your health problems?
  3. During the past seven days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study?
  4. During the past seven days, how many hours did you actually work?
  5. During the past seven days, how much did your health problems affect your productivity while you were working? (0-10, higher is more impact)
  6. During the past seven days, how much did your health problems affect your ability to do your regular daily activities, other than work at a job? By regular activities, we mean the usual activities you do, such as work around the house, shopping, childcare, exercising, studying, etc.(0-10, higher is more impact)
Change in quality of life | Baseline, 6, and 12 months
  Healthy Days Core Module (CDC HRQOL- 4)
  1. Would you say that in general your health is excellent, very good, good, fair or poor? Excellent Good Fair Poor
  2. Now thinking about your physical health, which includes physical illness and injury, how many days during the past 30 days was your physical health not good?
  3. Now thinking about your mental health, which includes stress, depression, and problems with emotions, how many days during the past 30 days was your mental health not good?
  4. During the past 30 days, approximately how many days did poor physical or mental health keep you from doing your usual activities, such as self-care, work, or recreation?

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Miller, MD, MPH, Principal Investigator — Stony Brook University Medical Center
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toro-Ramos T, Michaelides A, Anton M, Karim Z, Kang-Oh L, Argyrou C, Loukaidou E, Charitou MM, Sze W, Miller JD. Mobile Delivery of the Diabetes Prevention Program in People With Prediabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 8;8(7):e17842. doi: 10.2196/17842. PMID 32459631